CLINICAL TRIAL: NCT05703282
Title: A Parallel, Open-Label, Single-Dose Administration, Phase 1 Clinical Study to Assess the Safety and Pharmacokinetics of AD-104-A in Healthy Adult Volunteers and Patients With Renal Impairment
Brief Title: A Study to Assess the Safety and Pharmacokinetics of AD-104-A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AD-104PK_N
Record Dates: First submitted 2023-01-18; First posted 2023-01-30 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Renal Impairment 1 (Experimental): Test Drug: AD-104-A
  Interventions: Drug: AD-104-A
- Renal Impairment 2 (Experimental): Test Drug: AD-104-A
  Interventions: Drug: AD-104-A
- Renal Impairment 3 (Experimental): Test Drug: AD-104-A
  Interventions: Drug: AD-104-A
- Normal (Experimental): Test Drug: AD-104-A
  Interventions: Drug: AD-104-A

INTERVENTIONS:
Drug: AD-104-A — PO, Single-Dose, AD-104-A

SUMMARY:
Primary endpoint of this study is to evaluate the pharmacokinetic characteristics of AD-104-A

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the pharmacokinetic characteristics of AD-104-A in Healthy Adult Volunteers and Patients with Renal Impairment

ELIGIBILITY:
Inclusion Criteria:

For all subjects

* Adults aged 19 years and older
* Body mass index(BMI) of 18 to 30 kg/m2
* Voluntarily given written informed consent

For renal Impairment subjects

* 30 ≤ eGFR < 90 mL/min/1.73m^2

For healthy subjects

* eGFR ≥ 90 mL/min/1.73m^2

Exclusion Criteria:

* Participation in another clinical study with an investigational drug within the 6 months from scheduled first administration
* Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Cmax | pre-dose to 192 hours
  To assess the Cmax of AD-104-A
AUC | pre-dose to 192 hours
  To assess the AUC of AD-104-A

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea